CLINICAL TRIAL: NCT05900700
Title: An Open-Label Study of the Feasibility and Usability of a Digital Psychoeducational Social Network Intervention for Suicidal Adolescents
Brief Title: Digital Youth-Nominated Support Team (YST) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alejandra Arango, Assistant Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00221931; 5R43MH128431-02 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Suicide
Keywords: Social network; Website
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eYST website (Experimental)
  Interventions: Behavioral: eYST website

INTERVENTIONS:
Behavioral: eYST website — The website is a psychoeducational, social support program for adolescents at risk for suicide

SUMMARY:
The Electronic Youth-Nominated Support Team (eYST), is experimental. The purpose of this study is to get feedback from users about eYST. Another purpose of this study is to learn how well eYST helps youth.

DETAILED DESCRIPTION:
Assessment data from multiple stakeholders (i.e., youth, parents, and support adults) will be collected at baseline, 4 weeks, 8 weeks, and 12 weeks via self-report and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient psychiatric patients who have attempted suicide or have documented Suicide ideation (SI) and a plan to harm themselves at admission.
2. Understand written and spoken English.
3. Own a smartphone or mobile phone.
4. Willing and able to complete enrollment procedures.
5. Parent or guardian and youth able to understand the nature of the study and provide written informed consent and assent for youth
6. Patients who are able to provide at least one verifiable contact for emergency or tracking purposes.

Exclusion Criteria:

1. Patients with active psychosis.
2. Patients experiencing substance withdrawal.
3. Currently enrolled in other treatment studies for the symptoms and behaviors targeted.
4. Patient unwilling or unable to wear a mask during in person study procedures, if mandated due to current COVID/health safety guidelines.
5. Patients who in the judgment of the investigator would have an unfavorable risk or benefit profile with respect to eYST.
6. Any other psychiatric or medical condition or custody arrangement that in the investigators' opinion would preclude informed consent or assent or participation in the trial.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) score System Usability Scale (SUS) | Up to week 14
  10-item measure. Scores range from 0 to 100. The researchers will calculate the mean score. A mean score of 68 is the minimal indicator of usability.
Frequency of use of app | Up to week 12
  Frequency of eYST platform use will be tracked for each participant user. The researchers will record the number of logins.
Duration of use of app | Up to week 12
  The researchers will record the duration of app use.

SECONDARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Up to week 14
  Items are scored on a 5-point scale ranging from 1 to 5 (completely disagree to completely agree). Higher scores indicated higher perceived intervention feasibility.
Acceptability of Intervention Measure (AIM) | Up to week 14
  Items are scored on a 5-point scale ranging from 1 to 5 (completely disagree to completely agree). Higher scores indicate higher acceptability.
Intervention Appropriateness Measure (IAM) | Up to week 14
  Items are scored on a 5-point scale ranging from 1 to 5 (completely disagree to completely agree). Higher scores indicate higher perceived intervention appropriateness.
Client Satisfaction Questionnaire (CSQ-I) | Up to week 14
  The CSQ-I is a valid and reliable scale for measuring overall satisfaction with health and human services, including digital or internet-based intervention. This will be adapted for use with youth, parents and support adults. The adapted scales each have 8 items in a likert scale ranging from 8-32 where higher numbers indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Arango, Principal Investigator — University of Michigan; Patricia Simon, Study Director — Oui Therapeutics, Inc.
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT05900700/Prot_SAP_001.pdf
  • Informed Consent Form (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT05900700/ICF_000.pdf